CLINICAL TRIAL: NCT06918847
Title: Comparative Effectiveness of Myofacial Release vs Cupping Therapy on Quality of Life in Restless Leg Syndrome With Knee O.A.A RCT
Brief Title: Comparative Effectiveness of Myofacial Release vs Cupping Therapy on Quality of Life in Restless Leg Syndrome With Knee O.A.
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tooba Batool, Principal investigator, a Physiotherapist, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3866
Record Dates: First submitted 2025-04-08; First posted 2025-04-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Restless Leg Syndrome With Knee OA; Sleep Disorder
Keywords: Restless leg syndrome; knee OA; cupping therapy; myofacial release
MeSH Terms: conditions — Sleep Wake Disorders; Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A will be given treatment with myofacial release (Experimental): Myofascial release (MFR) for the calf muscle will be administered with the patient in a prone position, holding for 120 seconds. The Myofacial release technique involves allowing the lateral aspect of the therapist's thumb to sink into the central portion of the muscle belly. Myofacial release will be performed for 15 minutes.
  Interventions: Other: Myofacial release
- Group B will be given treatment with dynamic cupping therapy (Experimental): In dynamic cupping therapy, patients will be comfortably positioned in a prone position, ensuring that the lower limb is exposed and accessible for treatment. Appropriately sized cups will be selected and applied to the calf and hamstrings region. Prior to application, a small amount of lubricant or oil will be applied to facilitate the smooth movement of the cups over the skin surface during the therapy. The technique of dynamic cupping will involve compressing the cups and gently situating them onto the area being treated, applying the necessary force to generate negative pressure. The duration of dynamic cupping therapy will be 10 minutes.
  Interventions: Other: Dynamic cupping therapy

INTERVENTIONS:
Other: Myofacial release — Myofascial release (MFR) for the calf muscle will be administered with the patient in a prone position, holding for 120 seconds. The MFR technique involves allowing the lateral aspect of the therapist's thumb to sink into the central portion of the muscle belly. MFR will be performed for 15 minutes.
  Other Names: MFR
  Arms: Group A will be given treatment with myofacial release
Other: Dynamic cupping therapy — In dynamic cupping therapy, patients will be comfortably positioned in a prone position, ensuring that the lower limb is exposed and accessible for treatment. Appropriately sized cups will be selected and applied to the calf and hamstrings region. Prior to application, a small amount of lubricant or oil will be applied to facilitate the smooth movement of the cups over the skin surface during the therapy. The technique of dynamic cupping will involve compressing the cups and gently situating them onto the area being treated, applying the necessary force to generate negative pressure. The duration of dynamic cupping therapy will be 10 minutes.
  Arms: Group B will be given treatment with dynamic cupping therapy

SUMMARY:
The aim of this study is to determine effectiveness of Myofascial Release and Cupping Therapy on Quality of Life in Restless Leg Syndrome with knee Osteoarthritis. Holding this aim, a Randomized control trial will be conducted at physiotherapy out patient department of Dow Institute of Physical Medicine and Rehabilitation.

The subjects will first be screened by the principal investigator, physiotherapist, using the criteria of International Restless Leg Syndrome Study Group (IRLSSG). Each selected subject will go for random allocation in one of the two treatment groups with different interventions with the help of a computer-generated randomization sheet. The group A will be provided with myofacial release whereas the group B will receive cupping therapy while cryotherapy and passive lower limb stretches (hamstring and calf muscles) will be applied to both the groups as standard treatment. Assessment will be done at baseline and will re-evaluate at the post intervention session through an assessment form. Physical therapist but not the principal investigator will assess who will be unaware to the type of intervention administered.

Outcome measures will be Pittsburgh sleep quality index, Visual Analog Scale for pain assessment, Restless leg syndrome Quality of life questionnaire (RLS-QOL), International Restless leg syndrome Study Group Rating Scale (IRLSSG RS) and passive straight leg raise (PSLR). Total 12 sessions will be given for duration of 4weeks on alternate days.

ELIGIBILITY:
Inclusion Criteria:

1. grade 2, 3 and 4 knee OA by the Kellgren Lawrence classification
2. Bilateral or unilateral both knee OA
3. Age 40 to 70 years
4. Patients who were meeting the International Restless Leg Syndrome Study Group (IRLSSG) eligibility criteria

Exclusion Criteria:

1. patients with cognitive dysfunction
2. Rheumatoid arthritis
3. patients with neurological disorders
4. Medical conditions covering (cardiovascular disease, neurological disorders, severe psychiatric illness or pregnancy)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Restless leg syndrome quality of life Questionnaire | Assessment of outcome measure will be done at baseline and at the post intervention i.e 4 weeks.
  The Restless Leg Syndrome Quality of Life Questionnaire is a scale ranges from 0-100 with a desirable internal consistency (Cronbach's alpha =0.92) and test-retest reliability (intraclass correlation coefficient=0.84.All items possess considerable convergent validity.
International restless leg syndrome study group rating scale | Assessment of outcome measure will be done at baseline and at the post intervention i.e 4 weeks.
  The International restless leg syndrome study group rating scale comprises of 10 questions with ratings 0 to 4. The scale is a face-to-face interview validated questionnaire to clear the ambiguities of the subjects regarding the questions given.
  IRLSSG RS Inter rater reliability ICC = 0.97 IRLSSG RS Test-retest reliability ICC = 0.87 Internal consistency (cronbach's alpha) = 0.95 Criterion validity = 0.73.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guo S, Huang J, Jiang H, Han C, Li J, Xu X, Zhang G, Lin Z, Xiong N, Wang T. Restless Legs Syndrome: From Pathophysiology to Clinical Diagnosis and Management. Front Aging Neurosci. 2017 Jun 2;9:171. doi: 10.3389/fnagi.2017.00171. eCollection 2017. PMID 28626420
- [Result] Vlasie A, Trifu SC, Lupuleac C, Kohn B, Cristea MB. Restless legs syndrome: An overview of pathophysiology, comorbidities and therapeutic approaches (Review). Exp Ther Med. 2022 Feb;23(2):185. doi: 10.3892/etm.2021.11108. Epub 2021 Dec 30. PMID 35069866
- See also: Exploration of restless legs syndrome under the new concept: A review — https://journals.lww.com/md-journal/fulltext/2022/12160/exploration_of_restless_legs_syndrome_under_the.45